CLINICAL TRIAL: NCT03409731
Title: Absorb GT1 Bioresorbable Vascular Scaffold (BVS) System Post-marketing Surveillance (PMS)
Brief Title: Absorb GT1 Japan PMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 16-310
Record Dates: First submitted 2017-05-18; First posted 2018-01-24 (Actual); Results first posted 2019-01-03 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-05

CONDITIONS: Ischemic Heart Disease; Angina Pectoris; Coronary Artery Disease; Coronary Artery Occlusion; Myocardial Ischemia
Keywords: Drug eluting Bio-resolvable Scaffold (BRS); Bio-resolvable Scaffold (BRS); Real world
MeSH Terms: conditions — Myocardial Ischemia; Angina Pectoris; Coronary Artery Disease; Coronary Occlusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Absorb GT1 BVS (Other): Patients receiving Absorb GT1 Bioresorbable Vascular Scaffold System.
  Interventions: Device: ABSORB GT1 BVS

INTERVENTIONS:
Device: ABSORB GT1 BVS — Patients receiving Absorb GT1 BVS

SUMMARY:
The purpose of the Surveillance is to know the frequency and status of adverse device effects and adverse events in order to assure the safety of the new medical device, and to collect efficacy and safety information for evaluating clinical use results.

ELIGIBILITY:
Inclusion Criteria:

* General Percutaneous coronary intervention (PCI) population.

Exclusion Criteria:

* No specific exclusion criteria.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2016-12-13 (Actual); Primary Completion 2023-02-06 (Actual); Study Completion 2023-02-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Masato Nakamura, MD, Principal Investigator — Toho University Ohashi Medical Hospital
Locations (15):
- Japan (15):
  - Nagoya Daini Red Cross Hospital, Nagoya, Aichi-ken
  - Shin Tokyo Hospital, Matsudo, Chiba
  - Shin Koga Hospital, Kurume, Fukuoka
  - Hanaoka Seishu Memorial Cardiovascular Clinic, Sapporo, Hokkaido
  - Kobe University, Kobe, Hyōgo
  - Iwate Medical University, Morioka, Iwate
  - Shonan Kamakura General Hospital, Kamakura, Kanagawa
  - Kurashiki Central Hospital, Kurashiki, Okayama-ken
  - Saitama Sekishinkai Hospital, Sayama, Saitama
  - Mitsui Memorial Museum, Chiyoda City, Tokyo
  - Toho University Ohashi Medical Center, Meguro City, Tokyo
  - Teikyo University, tabashi City, Tokyo
  - Saiseikai Kumamoto Hospital, Kumamoto
  - Miyazaki Medical Association Hospital, Miyazaki
  - Sakurabashi Watanabe Hospital, Osaka

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Nakamura M, Suzuki N, Fujii K, Furuya J, Kawasaki T, Kimura T, Sakamoto T, Tanabe K, Kusano H, Stockelman KA, Kozuma K. The Absorb GT1 Bioresorbable Vascular Scaffold System - 5-Year Post-Market Surveillance Study in Japan. Circ J. 2024 May 24;88(6):863-872. doi: 10.1253/circj.CJ-23-0877. Epub 2024 Mar 13. PMID 38479861

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This surveillance planned to consecutively enroll two thousand (2,000) patients. However, in September 2017, Abbott Vascular decided to stop selling the Absorb GT1 system globally, as result of low commercial sales uptake compared to the prediction. Surveillance sites could continue to use the device and register patients until December 15, 2017. As a result, 135 patients were enrolled (treatment with Absorb GT1 attempted, i.e., ITT) by December 11, 2017.
Period: Overall Study
Arm/Group | Absorb GT1 BVS
Started | 135
Completed | 114
Not Completed | 21
Not completed — Withdrawal by Subject | 17
Not completed — Death | 4

BASELINE CHARACTERISTICS:
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 135
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The number of participants analyzed includes subjects who had available follow-up data at that time frame. The analysis excludes subjects who are truly lost to follow-up
  years | 64.0 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 114
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 135
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 135
Region of Enrollment [Number; unit: participants]
  Japan | 135
Diabetes Mellitus [Count of Participants; unit: Participants] | 53
Dyslipidemia [Count of Participants; unit: Participants] | 84
Hypertension [Count of Participants; unit: Participants] | 93
Renal Failure [Count of Participants; unit: Participants] | 5
Prior Coronary Intervention [Count of Participants; unit: Participants] | 35
Previous Myocardial Infarction (MI) [Count of Participants; unit: Participants] | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Acute Scaffold Thrombosis (ST)
Description: Criteria: ST rate (in 2,000 patients : sum of Phase 1 and Phase 2), Success Criteria: ST rate at 3 months is ≤ 18 patients (0.9%).
  Scaffold/Stent thrombosis should be reported as a cumulative value at the different time points and with the different separate time points. Time 0 is defined as the time point after the guiding catheter has been removed and the subject left the catheterization lab.
  Timings:
  Acute scaffold/stent thrombosis : 0 - 24 hours post stent implantation; Subacute scaffold/stent thrombosis: >24 hours - 30 days post stent implantation; Late scaffold/stent thrombosis: 30 days - 1 year post stent implantation; Very late scaffold/stent thrombosis: >1 year post stent implantation.
Time Frame: Day 0
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Number; unit: participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 134
participants
  Definite | 0
  Probable | 0
  Definite/Probable | 0

2. Primary Outcome: Number of Participants With Sub Acute Scaffold Thrombosis (ST)
Description: Criteria: ST rate (in 2,000 patients : sum of Phase 1 and Phase 2), Success Criteria: ST rate at 3 months is ≤ 18 patients (0.9%).
  Scaffold/Stent thrombosis should be reported as a cumulative value at the different time points and with the different separate time points. Time 0 is defined as the time point after the guiding catheter has been removed and the subject left the catheterization lab.
  Timings:
  Acute scaffold/stent thrombosis : 0 - 24 hours post stent implantation Subacute scaffold/stent thrombosis: >24 hours - 30 days post stent implantation Late scaffold/stent thrombosis: 30 days - 1 year post stent implantation Very late scaffold/stent thrombosis: >1 year post stent implantation.
Time Frame: >1 to 30 days
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Number; unit: participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 134
participants
  Definite | 0
  Probable | 0
  Definite/Probable | 0

3. Primary Outcome: Number of Participants With Late Scaffold Thrombosis (ST)
Description: Criteria: ST rate (in 2,000 patients : sum of Phase 1 and Phase 2),Success Criteria: ST rate at 3 months is ≤ 18 patients (0.9%). Scaffold/Stent thrombosis should be reported as a cumulative value at the different time points and with the different separate time points. Time 0 is defined as the time point after the guiding catheter has been removed and the subject left the catheterization lab.
  Timings:
  Acute scaffold/stent thrombosis : 0 - 24 hours post stent implantation Subacute scaffold/stent thrombosis: >24 hours - 30 days post stent implantation Late scaffold/stent thrombosis: 30 days - 1 year post stent implantation Very late scaffold/stent thrombosis: >1 year post stent implantation.
Time Frame: 31 to 90 days
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Number; unit: participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 134
participants
  Definite | 0
  Probable | 0
  Definite/Probable | 0

4. Primary Outcome: Number of Participants With Late Scaffold Thrombosis (ST)
Description: as for outcome 3
Time Frame: 31 to 365 days
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Number; unit: participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 134
participants
  Definite | 0
  Probable | 0
  Definite/Probable | 0

5. Primary Outcome: Number of Participants With Very Late Scaffold Thrombosis (ST)
Description: Criteria: ST rate (in 2,000 patients : sum of Phase 1 and Phase 2),Success Criteria: ST rate at 3 months is ≤ 18 patients (0.9%). Scaffold/Stent thrombosis should be reported as a cumulative value at the different time points and with the different separate time points. Time 0 is defined as the time point after the guiding catheter has been removed and the subject left the catheterization lab.
  Timings:
  Acute scaffold/stent thrombosis : 0 - 24 hours post stent implantation; Subacute scaffold/stent thrombosis: >24 hours - 30 days post stent implantation; Late scaffold/stent thrombosis: 30 days - 1 year post stent implantation; Very late scaffold/stent thrombosis: >1 year post stent implantation.
Time Frame: 366 to 730 days
Population: The number of participants analyzed includes subjects who had available follow-up data at that time frame. The analysis excludes subjects who are truly lost to follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 130
Participants
  Definite | 0
  Probable | 0
  Definite/Probable | 0

6. Primary Outcome: Number of Participants With Overall Scaffold Thrombosis (ST)
Description: as for outcome 5
Time Frame: 0 to 90 days
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 134
Participants
  Definite | 0
  Probable | 0
  Definite/Probable | 0

7. Primary Outcome: Number of Participants With Cumulative Scaffold Thrombosis
Description: as for outcome 2
Time Frame: 0 to 90 days
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Number; unit: participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 134
participants
  Definite | 0
  Probable | 0
  Definite/Probable | 0

8. Primary Outcome: Number of Participants With Cumulative Scaffold Thrombosis
Description: as for outcome 2
Time Frame: 0 to 730 days
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 131
Participants
  Definite | 0
  Probable | 0
  Definite/Probable | 0

9. Primary Outcome: Number of Participants With Exclusion of Very Small Vessels
Description: For Phase 1 patients, Angiograms and IVUS/OCT images taken during procedure will be sent immediately to the core lab. Additional training or revision of registration criteria may occur as required in order to exclude almost all lesions with RVD < 2.5 mm from registration by the last half of Phase 1.
Time Frame: During index procedure, "54.8 ± 27.6 min"
Population: Full Analysis Set (phase 1 participants with Absorb GT1)
Measure: Number; unit: participants
Units Other Than Participants: Lesions
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 135
Number analyzed (Lesions) | 139
participants
  < 2.25 mm | 18
  ≥ 2.25 mm - < 2.5 mm | 26
  ≥ 2.5 mm - ≤ 3.5 mm | 91
  > 3.5 mm | 4

10. Primary Outcome: Number of Participants With Scaffold Apposition Assessed by Intravascular Imaging
Description: IVUS/OCT images taken during procedure will be sent immediately to the core lab, which will analyze the images and give feedback to the site as required. Images of ST, if occurred, will also be sent to the core lab.
Time Frame: During index procedure, "54.8 ± 27.6 min"
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 135
Participants | 5

11. Primary Outcome: Number of Participants With Composite of Device Deficiencies
Description: Device deficiencies: Number of participants with at least one of the following Device deficiencies
  1. Lesion/implant failure
  2. Delivery difficulty (finally delivered)
  3. Re-crossing failure
  4. Re-crossing difficulty
  5. Post-dilatation balloon
  6. Optical Coherence Tomography (OCT)/Intravascular Ultrasound (IVUS)
  7. Instruction for Use (IFU) not included
  8. Major Strut Malapposition
  9. Strut Fracture within 6 months
Time Frame: During index procedure, "54.8 ± 27.6 min"
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 135
Participants
  Lesion/implant failure | 0
  Delivery difficulty (finally delivered) | 6
  Re-crossing failure | 1
  Re-crossing difficulty | 0
  Post-dilatation balloon+OCT/IVUS | 11
  IFU not included | 1
  Major Strut Malapposition | 1
  Strut Fracture within 6 months | 1

12. Primary Outcome: Number of Participants With Late Scaffold Thrombosis (ST)
Description: Criteria: ST rate (in 2,000 patients: sum of Phase 1 and Phase2), Success Criteria: ST rate at 3 months is ≤ 18 patients (0.9%). Scaffold/Stent thrombosis should be reported as a cumulative value at the different time points and with the different separate time points. Time 0 is defined as the time point after the guiding catheter has been removed and the subject left the catheterization lab.
  Timings: Acute scaffold/stent thrombosis: 0 - 24 hours post stent implantation; Subacute scaffold/stent thrombosis: >24 hours - 30 days post stent implantation; Late scaffold/stent thrombosis: 30 days - 1 year post stent implantation; Very late scaffold/stent thrombosis: >1 year post stent implantation.
Time Frame: 731 - 1095 days
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 127
Participants
  Definite | 0
  Probable | 0
  Definite/Probable | 0

13. Primary Outcome: Number of Participants With Cumulative Scaffold Thrombosis
Description: as for outcome 5
Time Frame: 0 - 1095 days
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 128
Participants
  Definite | 0
  Probable | 0
  Definite/Probable | 0

14. Primary Outcome: Number of Participants With Very Late Scaffold Thrombosis (ST)
Description: as for outcome 5
Time Frame: 1096 - 1460 days
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 120
Participants
  Definite | 0
  Probable | 0
  Definite/Probable | 0

15. Primary Outcome: Number of Participants With Cumulative Scaffold Thrombosis
Description: as for outcome 5
Time Frame: 0 - 1460 days
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 122
Participants
  Definite | 0
  Probable | 0
  Definite/Probable | 0

16. Primary Outcome: Number of Participants With Cumulative Scaffold Thrombosis
Description: as for outcome 12
Time Frame: 0 - 1825 days
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Number; unit: participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 116
participants
  Definite | 0
  Probable | 0
  Definite/Probable | 0

17. Secondary Outcome: Number of All Death (Cardiac, Vascular, Non-Cardiovascular)
Description: Cardiac death: Any death due to proximate cardiac cause (e.g. MI, low-output failure, fatal arrhythmia), unwitnessed death and death of unknown cause, all procedure related deaths including those related to concomitant treatment.
  Vascular death: Death due to non-coronary vascular causes such as cerebrovascular disease, pulmonary embolism, ruptured aortic aneurysm, dissecting aneurysm, or other vascular cause.
  Non-cardiovascular death: Any death not covered by the above definitions such as death caused by infection, malignancy, sepsis, pulmonary causes, accident, suicide or trauma.
Time Frame: 0 to 30 days
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 134
Participants | 0

18. Secondary Outcome: Number of All Death (Cardiac, Vascular, Non-Cardiovascular)
Description: as for outcome 17
Time Frame: 0 to 90 days
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 134
Participants | 0

19. Secondary Outcome: Number of All Death (Cardiac, Vascular, Non-Cardiovascular)
Description: as for outcome 17
Time Frame: 0 to 1 year
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 134
Participants | 0

20. Secondary Outcome: Number of All Death (Cardiac, Vascular, Non-Cardiovascular)
Description: as for outcome 17
Time Frame: 0 to 2 years
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 131
Participants | 2

21. Secondary Outcome: Number of Participants With All Myocardial Infarction (MI)
Description: Myocardial Infarction (MI) - Q wave MI: Development of new, pathological Q wave on the ECG.
  All myocardial infarction includes target vessel myocardial infarction (TV-MI) and not attributable to target vessel myocardial infarction (NTV-MI)
Time Frame: 0 to 30 days
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 134
Participants | 0

22. Secondary Outcome: Number of Participants With All Myocardial Infarction (MI)
Description: as for outcome 21
Time Frame: 0 to 90 days
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 134
Participants | 0

23. Secondary Outcome: Number of Participants With All Myocardial Infarction (MI)
Description: as for outcome 21
Time Frame: 0 to 1 year
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 134
Participants | 0

24. Secondary Outcome: Number of Participants With All Myocardial Infarction (MI)
Description: as for outcome 21
Time Frame: 0 to 2 years
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 131
Participants | 0

25. Secondary Outcome: Number of Participants With All Target Lesion Revascularization (TLR)
Description: Target Lesion Revascularization is defined as any repeat percutaneous intervention of the target lesion or bypass surgery of the target vessel performed for restenosis or other complication of the target lesion. All TLR should be classified prospectively as clinically indicated [CI] or not clinically indicated by the investigator prior to repeat angiography. An independent angiographic core laboratory should verify that the severity of percent diameter stenosis meets requirements for clinical indication and will overrule in cases where investigator reports are not in agreement.
  The target lesion is defined as the treated segment from 5 mm proximal to the stent and to 5 mm distal to the scaffold/stent.
Time Frame: 0 to 30 days
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 134
Participants | 1

26. Secondary Outcome: Number of Participants With All Target Lesion Revascularization (TLR)
Description: as for outcome 25
Time Frame: 0 to 90 days
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 134
Participants | 1

27. Secondary Outcome: Number of Participants With All Target Lesion Revascularization (TLR)
Description: as for outcome 25
Time Frame: 0 to 1 year
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 134
Participants | 1

28. Secondary Outcome: Number of Participants With All Target Lesion Revascularization (TLR)
Description: as for outcome 25
Time Frame: 0 to 2 years
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 131
Participants | 3

29. Secondary Outcome: Number of Participants With All Target Vessel Revascularization (TVR)
Description: Target Vessel Revascularization (TVR) is defined as any repeat percutaneous intervention or surgical bypass of any segment of the target vessel. The target vessel is defined as the entire major coronary vessel proximal and distal to the target lesion which includes upstream and downstream branches and the target lesion itself.
Time Frame: 0 to 30 days
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 134
Participants | 1

30. Secondary Outcome: Number of Participants With All Target Vessel Revascularization (TVR)
Description: as for outcome 29
Time Frame: 0 to 90 days
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 134
Participants | 1

31. Secondary Outcome: Number of Participants With All Target Vessel Revascularization (TVR)
Description: as for outcome 29
Time Frame: 0 to 1 year
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 134
Participants | 1

32. Secondary Outcome: Number of Participants With All Target Vessel Revascularization (TVR)
Description: as for outcome 29
Time Frame: 0 to 2 years
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 131
Participants | 4

33. Secondary Outcome: Number of Participants With All Coronary Revascularization
Description: All coronary revascularization is a composite of coronary artery bypass grafting (CABG) and percutaneous coronary intervention (PCI)
Time Frame: 0 to 30 days
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 134
Participants | 1

34. Secondary Outcome: Number of Participants With All Coronary Revascularization
Description: as for outcome 33
Time Frame: 0 to 90 days
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 134
Participants | 1

35. Secondary Outcome: Number of Participants With All Coronary Revascularization
Description: as for outcome 33
Time Frame: 0 to 1 year
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 134
Participants | 3

36. Secondary Outcome: Number of Participants With All Coronary Revascularization
Description: as for outcome 33
Time Frame: 0 to 2 years
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 131
Participants | 9

37. Secondary Outcome: Number of Death/MI/All Revascularization (DMR)
Description: DMR is the composite of All Death, All Myocardial infarction (MI) and All Revascularization
Time Frame: 0 to 30 days
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 134
Participants | 1

38. Secondary Outcome: Number of Death/MI/All Revascularization (DMR)
Description: DMR is the composite of All Death, All Myocardial infarction (MI) and All Revascularization
Time Frame: 0 to 90 days
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 134
Participants | 1

39. Secondary Outcome: Number of Death/MI/All Revascularization (DMR)
Description: DMR is the composite of All Death, All Myocardial infarction (MI) and All Revascularization
Time Frame: 0 to 1 year
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 134
Participants | 3

40. Secondary Outcome: Number of Death/MI/All Revascularization (DMR)
Description: DMR is the composite of All Death, All Myocardial infarction (MI) and All Revascularization
Time Frame: 0 to 2 years
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 131
Participants | 11

41. Secondary Outcome: Number of Participants With Target Vessel Failure (TVF)
Description: Target Vessel Failure (TVF) is the composite of Cardiac Death, Myocardial infarction (MI) or Ischemic-Driven Target Vessel Revascularization (ID-TVR).
Time Frame: 0 to 30 days
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 134
Participants | 0

42. Secondary Outcome: Number of Participants With Target Vessel Failure (TVF)
Description: as for outcome 41
Time Frame: 0 to 90 days
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 134
Participants | 0

43. Secondary Outcome: Number of Participants With Target Vessel Failure (TVF)
Description: as for outcome 41
Time Frame: 0 to 1 Year
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 134
Participants | 0

44. Secondary Outcome: Number of Participants With Target Vessel Failure (TVF)
Description: as for outcome 41
Time Frame: 0 to 2 years
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 131
Participants | 4

45. Secondary Outcome: Number of Major Adverse Cardiac Event (MACE)
Description: MACE is the composite of Cardiac death/All myocardial infarction (MI)/ Ischemia-driven Revascularization (ID-TLR)
Time Frame: 0 to 30 days
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 134
Participants | 0

46. Secondary Outcome: Number of Major Adverse Cardiac Event (MACE)
Description: MACE is the composite of Cardiac death/All myocardial infarction (MI)/ Ischemia-driven Revascularization (ID-TLR)
Time Frame: 0 to 90 days
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 134
Participants | 0

47. Secondary Outcome: Number of Major Adverse Cardiac Event (MACE)
Description: MACE is the composite of Cardiac death/All myocardial infarction (MI)/ Ischemia-driven Revascularization (ID-TLR)
Time Frame: 0 to 1 year
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 134
Participants | 0

48. Secondary Outcome: Number of Major Adverse Cardiac Event (MACE)
Description: MACE is the composite of Cardiac death/All myocardial infarction (MI)/ Ischemia-driven Revascularization (ID-TLR)
Time Frame: 0 to 2 years
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 131
Participants | 3

49. Secondary Outcome: Number of Cardiac Death/TV-MI/ID-TLR (TLF)
Description: Target Lesion Failure is composite of Cardiac death/ Target Vessel Myocardial Infarction (TV-MI)/ Ischemic-Driven Target Lesion Revascularization (ID-TLR).
Time Frame: 0 to 30 days
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 134
Participants | 0

50. Secondary Outcome: Number of Cardiac Death/TV-MI/ID-TLR (TLF)
Description: as for outcome 49
Time Frame: 0 to 90 days
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 134
Participants | 0

51. Secondary Outcome: Number of Cardiac Death/TV-MI/ID-TLR (TLF)
Description: as for outcome 49
Time Frame: 0 to 1 year
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 134
Participants | 0

52. Secondary Outcome: Number of Cardiac Death/TV-MI/ID-TLR (TLF)
Description: as for outcome 49
Time Frame: 0 to 2 years
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 131
Participants | 3

53. Secondary Outcome: Number of Participants With Cardiac Death/Myocardial Infarction (MI)
Description: Cardiac death: Any death due to proximate cardiac cause (e.g. MI, low-output failure, fatal arrhythmia), unwitnessed death and death of unknown cause, all procedure related deaths including those related to concomitant treatment.
Time Frame: 0 to 30 days
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 134
Participants | 0

54. Secondary Outcome: Number of Participants With Cardiac Death/Myocardial Infarction (MI)
Description: as for outcome 53
Time Frame: 0 to 90 days
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 134
Participants | 0

55. Secondary Outcome: Number of Participants With Cardiac Death/Myocardial Infarction (MI)
Description: as for outcome 53
Time Frame: 0 to 1 year
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 134
Participants | 0

56. Secondary Outcome: Number of Participants With Cardiac Death/Myocardial Infarction (MI)
Description: as for outcome 53
Time Frame: 0 to 2 years
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 131
Participants | 1

57. Secondary Outcome: Angiographic Endpoints (Core Lab Analysis): Lesion Morphology
Time Frame: Pre-procedure
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Number; unit: percentage of lesions
Units Other Than Participants: Lesions
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 135
Number analyzed (Lesions) | 139
percentage of lesions
  ACC/AHA Type B2/C | 51.8
  Severe/Moderate Calcification | 11.5
  Eccentric | 27.3
  Total Occlusion | 0.0

58. Secondary Outcome: Angiographic Endpoints (Core Lab Analysis):Thrombolysis in Myocardial Infarction (TIMI) Blood Flow
Description: TIMI 0 flow (no perfusion) refers to the absence of any antegrade flow beyond a coronary occlusion.
  TIMI 1 flow (penetration without perfusion) is faint antegrade coronary flow beyond the occlusion, with incomplete filling of the distal coronary bed.
  TIMI 2 flow (partial reperfusion) is delayed or sluggish antegrade flow with complete filling of the distal territory.
  TIMI 3 is normal flow which fills the distal coronary bed completely
Time Frame: Pre-procedure
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Number; unit: percentage of TIMI flow
Units Other Than Participants: Lesion
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 135
Number analyzed (Lesion) | 139
percentage of TIMI flow
  0 | 0.00
  1 | 0.72
  2 | 2.16
  3 | 97.12

59. Secondary Outcome: Angiographic Endpoints (Core Lab Analysis): Lesion Length
Description: Lesion Length (can be measured after successful post-dilatation)
Time Frame: Pre-procedure
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Lesions
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 135
Number analyzed (Lesions) | 139
mm | 13.84 (4.74)

60. Secondary Outcome: Angiographic Endpoints (Core Lab Analysis): Proximal Reference Vessel Diameter (RVD)
Description: Proximal RVD (can be measured after successful post-dilatation)
Time Frame: Pre-procedure
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Lesions
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 135
Number analyzed (Lesions) | 129
mm | 3.15 (0.49)

61. Secondary Outcome: Angiographic Endpoints (Core Lab Analysis): Distal RVD
Description: Distal RVD (can be measured after successful post-dilatation)
Time Frame: Pre-procedure
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Lesions
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 135
Number analyzed (Lesions) | 129
mm | 2.95 (0.39)

62. Secondary Outcome: Angiographic Endpoints (Core Lab Analysis): Minimum Lumen Diameter (MLD)
Description: Angiographic endpoint Minimum lumen diameter is defined as the shortest diameter through the center point of the lumen
Time Frame: Pre-procedure
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Lesions
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 135
Number analyzed (Lesions) | 139
mm | 1.00 (0.30)

63. Secondary Outcome: Angiographic Endpoints (Core Lab Analysis): Percent Diameter Stenosis (%DS)
Description: Percent Diameter Stenosis is defined as the value calculated as 100 * (1 - Minimum Luminal Diameter (MLD)/Reference vessel diameter (RVD)) using the mean values from two orthogonal views (when possible) by quantitative coronary angiography (QCA).
Time Frame: Pre-procedure
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Mean (Standard Deviation); unit: percentage of diameter
Units Other Than Participants: Lesions
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 135
Number analyzed (Lesions) | 139
percentage of diameter | 63.1 (9.5)

64. Secondary Outcome: Angiographic Endpoints (Core Lab Analysis): Thrombolysis in Myocardial Infarction (TIMI) Blood Flow
Description: as for outcome 58
Time Frame: Post-procedure (average procedure time of "54.8 ± 27.6 min")
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Number; unit: percentage of TIMI flow
Units Other Than Participants: Lesion
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 135
Number analyzed (Lesion) | 139
percentage of TIMI flow
  0 | 0.00
  1 | 0.72
  2 | 1.44
  3 | 97.84

65. Secondary Outcome: Angiographic Endpoints (Core Lab Analysis): MLD (In-segment)
Description: Angiographic endpoint. Minimum lumen diameter is defined as the shortest diameter through the center point of the lumen.
  In- Segment is defined as, within the margins of the stent or scaffold and 5 mm proximal and 5 mm distal to the stent or scaffold.
Time Frame: Post-procedure (average procedure time of "54.8 ± 27.6 min")
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Lesions
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 135
Number analyzed (Lesions) | 139
mm | 2.30 (0.38)

66. Secondary Outcome: Angiographic Endpoints (Core Lab Analysis): %DS (In-Segment )
Description: Percent Diameter Stenosis is defined as the value calculated as 100 * (1 - Minimum Luminal Diameter (MLD)/Reference vessel diameter (RVD)) using the mean values from two orthogonal views (when possible) by quantitative coronary angiography (QCA). In- Segment is defined as, within the margins of the stent or scaffold and 5 mm proximal and 5 mm distal to the stent or scaffold.
Time Frame: Post-procedure (average procedure time of "54.8 ± 27.6 min")
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Mean (Standard Deviation); unit: percentage of diameter
Units Other Than Participants: Lesions
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 135
Number analyzed (Lesions) | 139
percentage of diameter | 18.4 (6.3)

67. Secondary Outcome: Angiographic Endpoints (Core Lab Analysis): Acute Gain (In-Segment )
Description: The acute gain was defined as the difference between post- and pre procedural minimal lumen diameter (MLD).
Time Frame: Post-procedure (average procedure time of "54.8 ± 27.6 min")
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Lesions
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 135
Number analyzed (Lesions) | 139
mm | 1.29 (0.44)

68. Secondary Outcome: IVUS/OCT Endpoints (Core Lab Analysis): Lumen Diameter or Lumen Area (Proximal/Distal)
Time Frame: Pre-procedure (or after pre-dilatation)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mm^2
Units Other Than Participants: Lesions
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 135
Number analyzed (Lesions) | 139
mm^2
  Proximal | 8.04 (2.51)
  Distal | 6.29 (2.30)

69. Secondary Outcome: IVUS/OCT Endpoints (Core Lab Analysis): Lumen Diameter or Lumen Area (Proximal/Distal)
Time Frame: Post-procedure (average procedure time of "54.8 ± 27.6 min")
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Mean (Standard Deviation); unit: mm^2
Units Other Than Participants: Lesions
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 135
Number analyzed (Lesions) | 139
mm^2
  Proximal | 8.21 (2.47)
  Distal | 6.54 (2.21)

70. Secondary Outcome: IVUS/OCT Endpoints (Core Lab Analysis): Minimal Lumen Area
Time Frame: Post-procedure (average procedure time of "54.8 ± 27.6 min")
Population: Full Analysis Set (all participants with Absorb GT1).
Measure: Mean (Standard Deviation); unit: mm^2
Units Other Than Participants: Lesions
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 135
Number analyzed (Lesions) | 139
mm^2 | 6.86 (1.77)

71. Secondary Outcome: IVUS/OCT Endpoints (Core Lab Analysis): Percentage of Lesions With Strut Malapposition
Description: Percentage of lesions with strut malapposition will be calculated as mean ± standard deviation post-procedure
Time Frame: Post-procedure (average procedure time of "54.8 ± 27.6 min")
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Mean (Standard Deviation); unit: Percentage of lesions
Units Other Than Participants: Lesions
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 135
Number analyzed (Lesions) | 139
Percentage of lesions | 1.89 (3.63)

72. Secondary Outcome: IVUS/OCT Endpoints (Core Lab Analysis): Percentage of Strut Fracture
Description: Strut fracture will be measured as either number or percentage post-procedure
Time Frame: Post-procedure (average procedure time of "54.8 ± 27.6 min")
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Number; unit: Lesions
Units Other Than Participants: Lesions
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 135
Number analyzed (Lesions) | 139
Lesions
  Yes | 1
  No | 138

73. Secondary Outcome: Number of All Death (Cardiac, Vascular, Non-Cardiovascular)
Description: as for outcome 17
Time Frame: 3 years
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 129
Participants | 3

74. Secondary Outcome: Number of Participants With All Myocardial Infarction (MI)
Description: as for outcome 21
Time Frame: 3 years
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 129
Participants | 2

75. Secondary Outcome: Number of Participants With All Target Lesion Revascularization (TLR)
Description: as for outcome 25
Time Frame: 3 years
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 129
Participants | 4

76. Secondary Outcome: Number of Participants With All Target Vessel Revascularization (TVR)
Description: as for outcome 29
Time Frame: 3 years
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 129
Participants | 7

77. Secondary Outcome: Number of Participants With All Coronary Revascularization
Description: as for outcome 33
Time Frame: 3 years
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 129
Participants | 12

78. Secondary Outcome: Number of Death/MI/All Revascularization (DMR)
Description: DMR is the composite of All Death, All Myocardial infarction (MI) and All Revascularization
Time Frame: 3 years
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 129
Participants | 16

79. Secondary Outcome: Number of Participants With Target Vessel Failure (TVF)
Description: as for outcome 41
Time Frame: 3 years
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 129
Participants | 8

80. Secondary Outcome: Number of Major Adverse Cardiac Event (MACE)
Description: MACE is the composite of Cardiac death/All myocardial infarction (MI)/ Ischemia-driven Revascularization (ID-TLR)
Time Frame: 3 years
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 129
Participants | 6

81. Secondary Outcome: Number of Cardiac Death/TV-MI/ID-TLR (TLF)
Description: as for outcome 49
Time Frame: 3 years
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 129
Participants | 5

82. Secondary Outcome: Number of Participants With Cardiac Death/Myocardial Infarction (MI)
Description: as for outcome 53
Time Frame: 3 years
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 129
Participants | 3

83. Secondary Outcome: Number of All Death (Cardiac, Vascular, Non-Cardiovascular)
Description: as for outcome 17
Time Frame: 4 years
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 124
Participants | 4

84. Secondary Outcome: Number of Participants With All Myocardial Infarction (MI)
Description: as for outcome 21
Time Frame: 4 years
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 124
Participants | 2

85. Secondary Outcome: Number of Participants With All Target Lesion Revascularization (TLR)
Description: as for outcome 25
Time Frame: 4 years
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 124
Participants | 6

86. Secondary Outcome: Number of Participants With All Target Vessel Revascularization (TVR)
Description: as for outcome 29
Time Frame: 4 years
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 124
Participants | 11

87. Secondary Outcome: Number of Participants With All Coronary Revascularization
Description: as for outcome 33
Time Frame: 4 years
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 124
Participants | 16

88. Secondary Outcome: Number of Death/MI/All Revascularization (DMR)
Description: DMR is the composite of All Death, All Myocardial infarction (MI) and All Revascularization
Time Frame: 4 years
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 124
Participants | 22

89. Secondary Outcome: Number of Participants With Target Vessel Failure (TVF)
Description: as for outcome 41
Time Frame: 4 years
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 124
Participants | 11

90. Secondary Outcome: Number of Major Adverse Cardiac Event (MACE)
Description: MACE is the composite of Cardiac death/All myocardial infarction (MI)/ Ischemia-driven Revascularization (ID-TLR)
Time Frame: 4 years
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 124
Participants | 7

91. Secondary Outcome: Number of Cardiac Death/TV-MI/ID-TLR (TLF)
Description: as for outcome 49
Time Frame: 4 years
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 124
Participants | 6

92. Secondary Outcome: Number of Participants With Cardiac Death/Myocardial Infarction (MI)
Description: as for outcome 53
Time Frame: 4 years
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 124
Participants | 4

93. Secondary Outcome: Number of All Death (Cardiac, Vascular, Non-Cardiovascular)
Description: as for outcome 17
Time Frame: 5 years
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 118
Participants | 4

94. Secondary Outcome: Number of Participants With All Myocardial Infarction (MI)
Description: as for outcome 21
Time Frame: 5 years
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 118
Participants | 2

95. Secondary Outcome: Number of Participants With All Target Lesion Revascularization (TLR)
Description: as for outcome 25
Time Frame: 5 years
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 118
Participants | 6

96. Secondary Outcome: Number of Participants With All Target Vessel Revascularization (TVR)
Description: as for outcome 29
Time Frame: 5 years
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 118
Participants | 11

97. Secondary Outcome: Number of Death/MI/All Revascularization (DMR)
Description: DMR is the composite of All Death, All Myocardial infarction (MI) and All Revascularization.
Time Frame: 5 years
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 118
Participants | 23

98. Secondary Outcome: Number of Participants With Target Vessel Failure (TVF)
Description: as for outcome 41
Time Frame: 5 years
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 118
Participants | 11

99. Secondary Outcome: Number of Major Adverse Cardiac Event (MACE)
Description: MACE is the composite of Cardiac death/All myocardial infarction (MI)/ Ischemia-driven Revascularization (ID-TLR).
Time Frame: 5 years
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 118
Participants | 7

100. Secondary Outcome: Number of Cardiac Death/TV-MI/ID-TLR (TLF)
Description: as for outcome 49
Time Frame: 5 years
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 118
Participants | 6

101. Secondary Outcome: Number of Participants With Cardiac Death/Myocardial Infarction (MI)
Description: as for outcome 53
Time Frame: 5 years
Population: Full Analysis Set (all participants with Absorb GT1)
Measure: Count of Participants; unit: Participants
Arm/Group | Absorb GT1 BVS
Number analyzed (Participants) | 118
Participants | 4

ADVERSE EVENTS:
Time Frame: 5 Years
Arm/Group | Absorb GT1 BVS
All-Cause Mortality (participants affected / at risk) | 4/135
Serious Adverse Events (participants affected / at risk) | 43/135
Other Adverse Events (participants affected / at risk) | 8/135
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Absorb GT1 BVS (N=135)
Angina pectoris (Cardiac disorders) | 14
Angina, unstable (Cardiac disorders) | 2
Aortic valve stenosis (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 13
Myocardial infarction (Cardiac disorders) | 2
Sudden hearing loss (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Cataract (Eye disorders) | 2
Colitis ischaemic (Gastrointestinal disorders) | 2
Colonic polyp (Gastrointestinal disorders) | 3
Gastrointestinal inflammation (Gastrointestinal disorders) | 1
Sudden death (General disorders) | 1
Biliary colic (Hepatobiliary disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 2
Cholecystitis acute (Hepatobiliary disorders) | 1
Abdominal infection (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
Coronary artery restenosis (Injury, poisoning and procedural complications) | 2
Femur fracture (Injury, poisoning and procedural complications) | 1
In-stent coronary artery restenosis (Injury, poisoning and procedural complications) | 2
Pelvic fracture (Injury, poisoning and procedural complications) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Traumatic haematoma (Injury, poisoning and procedural complications) | 1
Traumatic lung injury (Injury, poisoning and procedural complications) | 1
Hepatic Enzyme Increased (Investigations) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Oesophageal Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Carotid artery stenosis (Nervous system disorders) | 2
Cerebral artery occlusion (Nervous system disorders) | 1
Hydrocephalus (Nervous system disorders) | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 1
Knee arthroplasty (Surgical and medical procedures) | 2
Aortic aneurysm (Vascular disorders) | 1
Haemorrhage (Vascular disorders) | 5
Subclavian artery stenosis (Vascular disorders) | 1
Phimosis (Congenital, familial and genetic disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Absorb GT1 BVS (N=135)
Coronary artery disease (Cardiac disorders) | 1
Thrombosis in Device (General disorders) | 1
Cerebral artery stenosis (Nervous system disorders) | 1
Dermal Eruption (Skin and subcutaneous tissue disorders) | 1
Coronary Revascularization (Surgical and medical procedures) | 1
Haemorrhage (Vascular disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2016-11-08): https://cdn.clinicaltrials.gov/large-docs/31/NCT03409731/Prot_002.pdf
  • Statistical Analysis Plan (2017-02-17): https://cdn.clinicaltrials.gov/large-docs/31/NCT03409731/SAP_003.pdf